CLINICAL TRIAL: NCT06394141
Title: MILESTONE: MobILe and tEchnological SoluTions for OccupatioNal drivErs
Brief Title: MILESTONE - MobILe and tEchnological SoluTions for OccupatioNal drivErs
Acronym: MILESTONE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Collaborators: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, An Neven, Associate Professor, Hasselt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MILESTONE; HBC.2021.0387 (Other Grant/Funding Number: Flanders Innovation & Entrepreneurship (VLAIO))
Record Dates: First submitted 2024-04-20; First posted 2024-05-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Healthy
Keywords: Occupational freight drivers; Stress reduction; Technological interventions

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Real-time triggers (Experimental): The first intervention group (n= 30 professional drivers) will receive real-time triggers related to acute stress and sleepiness/fatigue. The real-time feedback involves giving relevant triggers when exceeding some critical stress values or detecting events of 'energy-takers' based on accurate measurements of mental energy in a fully automated way. The selected triggers will be based on the co-creation workshops with drivers (e.g., auditive, visual) in order to select the most efficient (type or combination of) trigger(s) for the real-time feedback. The warning messages will be tailored to the preferences of the driver (e.g., personalized comfort- and safety-related settings) and aim to generate a warning message/signal meant to alert drivers and prevent they might end up with high stress levels.
  Interventions: Behavioral: Real-time triggers
- Personalized tailored feedback (Experimental): The second intervention group (n= 30 professional drivers) will receive personalized tailored feedback to reduce chronic stress and sleepiness/fatigue. The advice involves personalized (semi-)automatic feedback to drivers about a reduced stress level via the mobile app with automatic reports, as well as post-intervention during the next work break or at the end of the workday, based on the preferences of the driver. The (semi-)automatic feedback is based on the theory of Stages of Change, by which a driver will only receive relevant feedback based on their attitude and willingness during daily life.
  Interventions: Behavioral: Personalized tailored feedback
- Real-time triggers + Personalized tailored feedback (Experimental): The third intervention group (n= 30 professional drivers) will receive both real-time feedback related to acute stress and sleepiness/fatigue, as well as personalized tailored feedback related to chronic stress and sleepiness/fatigue, similar as in the first and second intervention groups.
  Interventions: Behavioral: Real-time triggers + Personalized tailored feedback
- App-supported exercise therapy (Experimental): The fourth intervention group (n= 30 professional drivers) will receive app-supported exercise therapy. The intervention will be based on principles of high-intensity training exercises that focus on the improvement of cardiorespiratory exercise capacity, as well as on the reduction of stress levels during work. Participants will receive instructions via the app to do some short, vigorous exercises adapted to their work environment at regular intervals, e.g., bending-and-stretching exercises with a weight in their hands, walking up and down the stairs of their vehicle for a few minutes, etc.
  Interventions: Behavioral: App-supported exercise therapy
- Conventional intervention (Active Comparator): The active control group (n= 20 professional drivers) will get a conventional intervention to reduce stress, e.g., mindfulness.
  Interventions: Behavioral: Conventional intervention
- Control group (No Intervention): The passive control group (n= 20 professional drivers) will get no intervention and will continue as normal without receiving any feedback.

INTERVENTIONS:
Behavioral: Real-time triggers — The first intervention group (n= 30 professional drivers) will receive real-time triggers related to acute stress and sleepiness/fatigue. The real-time feedback involves giving relevant triggers when exceeding some critical stress values or detecting events of 'energy-takers' based on accurate measurements of mental energy in a fully automated way. The selected triggers will be based on the co-creation workshops with drivers (e.g., auditive, visual) in order to select the most efficient (type or combination of) trigger(s) for the real-time feedback. The warning messages will be tailored to the preferences of the driver (e.g., personalized comfort- and safety-related settings) and aim to generate a warning message/signal meant to alert drivers and prevent they might end up with high stress levels
  Arms: Real-time triggers
Behavioral: Personalized tailored feedback — The second intervention group (n= 30 professional drivers) will receive personalized tailored feedback to reduce chronic stress and sleepiness/fatigue. The advice involves personalized (semi-)automatic feedback to drivers about a reduced stress level via the mobile app with automatic reports, as well as post-intervention during the next work break or at the end of the workday, based on the preferences of the driver. The (semi-)automatic feedback is based on the theory of Stages of Change, by which a driver will only receive relevant feedback based on their attitude and willingness during daily life.
  Arms: Personalized tailored feedback
Behavioral: Real-time triggers + Personalized tailored feedback — The third intervention group (n= 30 professional drivers) will receive both real-time feedback related to acute stress and sleepiness/fatigue, as well as personalized tailored feedback related to chronic stress and sleepiness/fatigue, similar as in the first and second intervention groups.
  Arms: Real-time triggers + Personalized tailored feedback
Behavioral: App-supported exercise therapy — The fourth intervention group (n= 30 professional drivers) will receive app-supported exercise therapy. The intervention will be based on principles of high-intensity training exercises that focus on the improvement of cardiorespiratory exercise capacity, as well as on the reduction of stress levels during work. Participants will receive instructions via the app to do some short, vigorous exercises adapted to their work environment at regular intervals, e.g., bending-and-stretching exercises with a weight in their hands, walking up and down the stairs of their vehicle for a few minutes, etc.
  Arms: App-supported exercise therapy
Behavioral: Conventional intervention — The active control group (n= 20 professional drivers) will get a conventional intervention to reduce stress, e.g., mindfulness.
  Arms: Conventional intervention

SUMMARY:
Professional drivers in freight transport often experience difficult, exhausting and stressful working conditions due to various reasons: irregular sleep patterns, uncertainty in traffic, frequently changing schedules, busy schedules, a lot of time away from home, etc. These working conditions can lead to significant health problems with a significant impact on road safety. According to the International Road Transport Union, Europe is currently facing the most acute driver shortage in decades; which threatens the continued growth of the road transport sector, and its ability to provide solutions to expected volume growth. Technology will play an important role in making road transport safer and more efficient. MILESTONE's overall objective is to develop and test technological interventions which are expected to reduce the difficult working conditions, stress, negative health effects of professional drivers.

DETAILED DESCRIPTION:
The overall objective of MILESTONE is to develop and test technological interventions to reduce the difficult working conditions, stress, negative health effects of professional drivers.

1. Understanding the impact of personal state and contextual stress on driving behavior and road safety, and aims to analyze the relationship between physiological and mental state (e.g., sleep quality, fatigue, sleepiness, stress, thermal comfort), general health status, work-related factors, external stressors, and driving parameters linked to road safety.
2. Developing an intervention to keep drivers within their "stress tolerance zone" (STZ) (personal zone within which stress is acceptable)
3. Analyzing the impact of the MILESTONE interventions for different categories of drivers (long-haul, short-haul and local delivery), compared to an active and passive control group

ELIGIBILITY:
Inclusion Criteria:

* Working as long-haul, short-haul, or local delivery driver (in a transport company or self-employed)
* Having a smartphone
* Dutch-speaking

Exclusion Criteria:

* No excessive alcohol use
* No drugs use
* Not having an infectious disease
* Not being pregnant

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Accumulated heart rate-based load measure (average of all trips during past 2 weeks) | At the beginning of the intervention, intermediate after 2 months (mid of intervention), at the end of the intervention after 4,5 months, and 3 months after the intervention (to measure the impact on a longer-term).
  Mental load (derived from the energy balance estimation, as an indication of stress), measured by accumulated heart rate-based load measure via wearable (average of all trips during past 2 weeks)

SECONDARY OUTCOMES:
Work Ability Index | At the beginning of the intervention, intermediate after 2 months (mid of intervention), at the end of the intervention after 4,5 months, and 3 months after the intervention (to measure the impact on a longer-term).
  A summary measure of 7 items (e.g., the demands of work, the worker's health status and resources) identifying the health risks and risks of early retirement. The final WAI score is calculated as the total unweighted score covering the WAI's seven dimensions, or indicators. The combination of dimension values results in a total WAI score that can range from 7 (unable to work) to 49 (full work ability).
36-item Short Form Healthy Survey | At the beginning of the intervention, intermediate after 2 months (mid of intervention), at the end of the intervention after 4,5 months, and 3 months after the intervention (to measure the impact on a longer-term).
  Measuring health-related quality of life, consisting of both a physical and mental component. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Perceived Stress Scale 10 | At the beginning of the intervention, intermediate after 2 months (mid of intervention), at the end of the intervention after 4,5 months, and 3 months after the intervention (to measure the impact on a longer-term).
  Measuring perceived stress. The questions ask about feelings and thoughts during the last month. In each case, respondents are asked how often they felt a certain way on a five-point scale from 'never' to 'very often'. Answers are then scored as follow: Never = 0; Almost never = 1; Sometimes = 2; Fairly often = 3; Very often = 4. To calculate a total PSS score, responses to the four positively stated items (items 4, 5, 7 and 8) first need to be reversed (i.e. 0 => 4; 1 => 3; 2 => 2; 3 => 1; 4 => 0). The PSS score is then obtained by summing across all items. Higher scores indicate higher levels of perceived stress.
Driving Behaviour Inventory - General Driver Stress | At the beginning of the intervention, intermediate after 2 months (mid of intervention), at the end of the intervention after 4,5 months, and 3 months after the intervention (to measure the impact on a longer-term).
  A 16-item instrument extracted from the Driver Behaviour Inventory that measures general driver stress. The DBI-Gen consists of 16 items that tap a general disposition, or "trait" susceptibility, to driver stress. Responses are made on a Likert scale ranging from 0 to 100, indicating the level of agreement with each statement. Scoring consisted of the mean response to the 16 tems, with higher scores indicating greater trait driver stress susceptibility.
General Self-Efficacy Scale | At the beginning of the intervention, intermediate after 2 months (mid of intervention), at the end of the intervention after 4,5 months, and 3 months after the intervention (to measure the impact on a longer-term).
  Measuring a broad and stable sense of personal competence to deal effectively with a variety of stressful situations. The total score is calculated by finding the sum of all 10 items. For the GSE, the total score ranges between 10 and 40, with a higher score indicating more self-efficacy.
Depression Anxiety Stress Scales | At the beginning of the intervention, intermediate after 2 months (mid of intervention), at the end of the intervention after 4,5 months, and 3 months after the intervention (to measure the impact on a longer-term).
  A 42-item self-report instrument designed to measure the related negative emotional states of depression, anxiety, tension/stress.The DASS assesses negative emotional symptoms by using a 4-point Likert scale, ranging from 0 to 3. It has 3 subscales (depression, anxiety, and stress) with 14 items in each subscale for the DASS 42. These subscales are scored by the addition of the total item scores, which can range from 0 to 42. Maximum score: 126 for the 42-item DASS. A higher score on the DASS indicates greater severity or frequency of these negative emotional symptoms.
Fatigue Assessment Scale | At the beginning of the intervention, intermediate after 2 months (mid of intervention), at the end of the intervention after 4,5 months, and 3 months after the intervention (to measure the impact on a longer-term).
  A short, valid, reliable and easy to administer unidimensional fatigue questionnaire. The FAS is a 10-item general fatigue questionnaire to assess fatigue. Five questions reflect physical fatigue and 5 questions (questions 3 and 6-9) mental fatigue. An answer to every question has to be given, even if the person does not have any complaints at the moment. Scores on question 4 and 10 should be recoded (1=5, 2=4, 3=3, 4=2, 5=1). Subsequently, the total FAS score can be calculated by summing the scores on all questions (recoded scores for questions 4 and 10). The total score ranges from 10 to 50. A total FAS score < 22 indicates no fatigue, a score ≥ 22 indicates fatigue.
Epworth Sleepiness Scale | At the beginning of the intervention, intermediate after 2 months (mid of intervention), at the end of the intervention after 4,5 months, and 3 months after the intervention (to measure the impact on a longer-term).
  To measure daytime sleepiness, asking the subject how likely he/she is to doze off or fall asleep in different situations of everyday life. The test is a list of eight situations in which the respondents rates his/her tendency to become sleepy on a scale of 0, no chance of dozing, to 3, high chance of dozing. All answers to the questions need to be added.The total score is based on a scale of 0 to 24, with a higher score means a higher respondent's sleepiness.

CONTACTS AND LOCATIONS:
Overall Officials: An Neven, PhD, Principal Investigator — Hasselt University - Transportation Research Institute (IMOB)
Locations (1):
- Hasselt University, Hasselt, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: No
GDPR

REFERENCES:
- See also: MILESTONE website — https://www.uhasselt.be/milestone